CLINICAL TRIAL: NCT01463202
Title: Effect of Timing of Postpartum Depot Medroxyprogesterone Acetate Administration on Breastfeeding Continuation, Contraceptive Continuation, and Postpartum Depression: a Randomized Trial
Brief Title: Timing of Postpartum Depot Medroxyprogesterone Acetate Administration on Breastfeeding, Contraceptive Continuation, and Depression
Acronym: DEPO-ABCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beatrice Chen (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor-Investigator, Beatrice Chen, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFP5-1
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Contraception; Postpartum Depression; Lactation
Keywords: Postpartum contraception; Contraceptive continuation; Breastfeeding; Postpartum depression; Progestins
MeSH Terms: conditions — Depression, Postpartum; Breast Feeding | interventions — N,N-dimethyl-4-anisidine; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMPA postpartum (Active Comparator): Depot medroxyprogesterone acetate postpartum
  Interventions: Drug: Depot medroxyprogesterone acetate
- DMPA at 4-6 weeks after delivery (Active Comparator): Depot medroxyprogesterone acetate at 4-6 weeks after delivery
  Interventions: Drug: Depot medroxyprogesterone acetate

INTERVENTIONS:
Drug: Depot medroxyprogesterone acetate — Postpartum administration of DMPA (prior to hospital discharge)
  Other Names: DMPA; Depo Provera
  Arms: DMPA postpartum
Drug: Depot medroxyprogesterone acetate — Delayed administration of DMPA (4-6 weeks postpartum)
  Other Names: DMPA; Depo Provera
  Arms: DMPA at 4-6 weeks after delivery

SUMMARY:
The investigators plan to enroll 184 women who are planning to breastfeed and use DMPA after delivery to find out whether the timing of postpartum administration of DMPA (prior to hospital discharge or 4-6 weeks after delivery) affects the duration or exclusivity of breastfeeding among women who plan to breastfeed their infants.

DETAILED DESCRIPTION:
In the United States, depot medroxyprogesterone acetate (DMPA) is given to women after delivery and before hospital discharge with the belief that women who delay starting DMPA may be more likely to become pregnant when they are not yet ready to be pregnant and that giving DMPA before discharge has little to no negative effect on breastfeeding. Administering DMPA to breastfeeding women has not been widely questioned because the limited existing studies do not show any adverse impact of DMPA on breastfeeding. However, these studies used inappropriate control groups and did not control for prior lactation experience.

The investigators plan to enroll 184 women who are planning to breastfeed and use DMPA after delivery to find out whether the timing of postpartum administration of DMPA (prior to hospital discharge or 4-6 weeks after delivery) affects the duration or exclusivity of breastfeeding among women who plan to breastfeed their infants. The investigators will also look at rates of use of highly effective contraception (defined as DMPA, intrauterine device, implant, sterilization, or lactational amenorrhea) and postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old and > 24 0/7 weeks pregnant at time of enrollment
* Planning to deliver at Magee-Womens Hospital and to breastfeed
* Plans to use DMPA for postpartum contraception for at least 6 months
* Willing and able to provide informed consent in English and to comply with study protocol

Exclusion Criteria:

* Intolerance of irregular vaginal bleeding
* Severe coagulation disorder
* Severe liver disease (LFTs >2x upper limits of normal at time of randomization)
* Contraindications to breastfeeding: maternal HIV infection; active herpes simplex with breast lesions; active varicella; active, untreated tuberculosis; antineoplastic, thyrotoxic, or immunosuppressive medications; concern that the infant may have galactosemia
* History of breast cancer, reduction or augmentation surgery
* History of severe clinical depression
* Multiple gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2011-11; Primary Completion 2017-02-13 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Coordinator, Principal Investigator — University of Pittsburgh
Locations (1):
- Center for Family Planning Research, Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Since participants could be recruited antepartum but may have changed their mind about breastfeeding or DMPA use post-partum, eligibility criteria were re-assessed postpartum, prior to randomization, thus the number of women enrolled in the study (184) does not equal the number of women randomized (157).
Period: Overall Study
Arm/Group | DMPA Postpartum | DMPA at 4-6 Weeks After Delivery
Started (27 ineligible postpartum (26 no longer eligible, 1 withdrew consent)) | 79 | 78
Completed | 79 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DMPA Postpartum | DMPA at 4-6 Weeks After Delivery | Total
Number analyzed (Participants) | 79 | 78 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (4.9) | 24.4 (4.7) | 24.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 78 | 157
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 9 | 20
  Black | 61 | 61 | 122
  Other | 7 | 8 | 15
  Hispanic | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Duration of Breastfeeding Among Women Who Plan to Breastfeed Their Infants After Postpartum or Delayed (4-6 Weeks Postpartum) Initiation of DMPA
Description: Any breastfeeding at specific time intervals postpartum
Time Frame: 2, 4, 6, 8 12, 16, 20, 24, and 28 weeks postpartum
Population: 1 ppt withdrawn postrandomization due to enrollment violation (did not meet eligibility criteria)
Measure: Count of Participants; unit: Participants
Arm/Group | DMPA Postpartum | DMPA at 4-6 Weeks After Delivery
Number analyzed (Participants) | 79 | 77
Participants
  2 weeks postpartum: Any breastfeeding | 71 | 70
  2 weeks postpartum: Formula only | 4 | 4
  2 weeks postpartum: Missed call | 4 | 3
  4 weeks postpartum: Any breastfeeding | 69 | 66
  4 weeks postpartum: Formula only | 4 | 7
  4 weeks postpartum: Missed call | 6 | 4
  6 weeks postpartum: Any breastfeeding | 61 | 63
  6 weeks postpartum: Formula only | 9 | 9
  6 weeks postpartum: Missed call | 9 | 5
  8 weeks postpartum: Any breastfeeding | 59 | 53
  8 weeks postpartum: Formula only | 14 | 16
  8 weeks postpartum: Missed call | 6 | 8
  12 weeks postpartum: number analyzed (Participants) | 79 | 76
  12 weeks postpartum: Any breastfeeding | 51 | 47
  12 weeks postpartum: Formula only | 22 | 21
  12 weeks postpartum: Missed call | 6 | 8
  16 weeks postpartum: number analyzed (Participants) | 78 | 76
  16 weeks postpartum: Any breastfeeding | 40 | 40
  16 weeks postpartum: Formula only | 30 | 28
  16 weeks postpartum: Missed call | 8 | 8
  20 weeks postpartum: number analyzed (Participants) | 78 | 76
  20 weeks postpartum: Any breastfeeding | 39 | 31
  20 weeks postpartum: Formula only | 29 | 34
  20 weeks postpartum: Missed call | 10 | 11
  24 weeks postpartum: number analyzed (Participants) | 78 | 76
  24 weeks postpartum: Any breastfeeding | 34 | 32
  24 weeks postpartum: Formula only | 32 | 34
  24 weeks postpartum: Missed call | 12 | 10
  28 weeks postpartum: number analyzed (Participants) | 78 | 76
  28 weeks postpartum: Any breastfeeding | 39 | 38
  28 weeks postpartum: Formula only | 28 | 25
  28 weeks postpartum: Missed call | 11 | 13

2. Secondary Outcome: Rates of Use of Highly Effective Contraception (Defined as DMPA, IUD, Implant, Sterilization, or Lactational Amenorrhea) After Postpartum or Delayed Initiation of DMPA
Description: Use of DMPA, IUD, implant, or sterilization
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DMPA Postpartum | DMPA at 4-6 Weeks After Delivery
Number analyzed (Participants) | 79 | 78
Participants
  DMPA, IUD, implant, or sterilization | 43 | 44
  Less effective than DMPA | 25 | 21
  Lost to followup | 11 | 13

3. Secondary Outcome: Rates of Postpartum Depression After Postpartum or Delayed Initiation of DMPA
Description: Edinburgh Postnatal Depression Scale (EPDS) score after postpartum or delayed initiation of DMPA: minimum possible score 0, maximum possible score 30; score of 12 or greater is a positive screen for postpartum depression
Time Frame: 8 weeks postpartum
Population: Excludes 14 participants with a missed call at 8 weeks postpartum
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | DMPA Postpartum | DMPA at 4-6 Weeks After Delivery
Number analyzed (Participants) | 73 | 69
scores on a scale | 1.0 [0 to 4] | 0 [0 to 5]

4. Secondary Outcome: Exclusivity of Breastfeeding Among Women Who Plan to Breastfeed Their Infants After Postpartum or Delayed (4-6 Weeks Postpartum) Initiation of DMPA
Description: Exclusive breastfeeding at specific time intervals postpartum
Time Frame: 2, 4, 6, 8, 12, 16, 20,24 and 28 weeks postpartum
Population: Two participants withdrew during follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | DMPA Postpartum | DMPA at 4-6 Weeks After Delivery
Number analyzed (Participants) | 79 | 77
Participants
  2 weeks postpartum: Exclusive breastfeeding | 38 | 37
  2 weeks postpartum: Any formula | 37 | 37
  2 weeks postpartum: Missed call | 4 | 3
  4 weeks postpartum: Exclusive breastfeeding | 29 | 28
  4 weeks postpartum: Any formula | 44 | 45
  4 weeks postpartum: Missed call | 6 | 4
  6 weeks postpartum: Exclusive breastfeeding | 25 | 25
  6 weeks postpartum: Any formula | 45 | 47
  6 weeks postpartum: Missed call | 9 | 5
  8 weeks postpartum: Exclusive breastfeeding | 23 | 19
  8 weeks postpartum: Any formula | 50 | 50
  8 weeks postpartum: Missed call | 6 | 8
  12 weeks postpartum: number analyzed (Participants) | 79 | 76
  12 weeks postpartum: Exclusive breastfeeding | 17 | 22
  12 weeks postpartum: Any formula | 56 | 46
  12 weeks postpartum: Missed call | 6 | 8
  16 weeks postpartum: number analyzed (Participants) | 78 | 76
  16 weeks postpartum: Exclusive breastfeeding | 13 | 15
  16 weeks postpartum: Any formula | 57 | 53
  16 weeks postpartum: Missed call | 8 | 8
  20 weeks postpartum: number analyzed (Participants) | 78 | 76
  20 weeks postpartum: Exclusive breastfeeding | 11 | 10
  20 weeks postpartum: Any formula | 57 | 55
  20 weeks postpartum: Missed call | 10 | 11
  24 weeks postpartum: number analyzed (Participants) | 78 | 76
  24 weeks postpartum: Exclusive breastfeeding | 9 | 10
  24 weeks postpartum: Any formula | 57 | 56
  24 weeks postpartum: Missed call | 12 | 10
  28 weeks postpartum: number analyzed (Participants) | 78 | 76
  28 weeks postpartum: Exclusive breastfeeding | 7 | 6
  28 weeks postpartum: Any formula | 60 | 57
  28 weeks postpartum: Missed call | 11 | 13

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | DMPA Postpartum | DMPA at 4-6 Weeks After Delivery
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/78
Other Adverse Events (participants affected / at risk) | 0/79 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT01463202/Prot_SAP_000.pdf